CLINICAL TRIAL: NCT00443937
Title: Pharmacokinetics of Everolimus and Enteric-Coated Mycophenolatesodium Before and After Withdrawal of Cyclosporine in Stable Renal Transplant Patients
Brief Title: Pharmacokinetics of Everolimus and Enteric-Coated Mycophenolatesodium Before and After Withdrawal of Cyclosporine in Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ADE05
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Renal Transplantation
Keywords: Kidney Transplantation; Renal Transplantation; Mycophenolate; Cyclosporine; Everolimus
MeSH Terms: interventions — Mycophenolic Acid; Everolimus

INTERVENTIONS:
Drug: enteric-coated mycophenolate sodium — oral
  Other Names: Myfortic
Drug: everolimus — oral
  Other Names: Certican

SUMMARY:
Cyclosporine (CNI), a potent immunosuppressive drug used in transplant recipients to prevent graft rejection, can cause renal impairment in some patients. The aims of this study are

* To determine the influence of CNI discontinuation on the drug exposure and key pharmacokinetic parameters of everolimus and enteric-coated mycophenolate sodium (EC-MPS)
* To determine the adequate dosing of everolimus and EC-MPS in a CNI-free regimen
* To investigate the CNI-free regimen with EC-MPS and everolimus with respect to safety (e.g. rejection rates) and tolerability
* To investigate renal function after CsA withdrawal

ELIGIBILITY:
Inclusion Criteria:

* Patients having a kidney transplant since at least 6 months but for no longer than 5 years.
* Patients in a stable condition in terms of graft function
* Patients currently receiving EC-MPS and CsA with or without corticosteroids as part of their immunosuppressive regimen for at least 1 month prior to Baseline
* Females of childbearing potential must have a negative serum pregnancy test prior to study inclusion. If positive, the patient will not be enrolled. Effective contraception must be used during the trial.

Exclusion Criteria:

* Patients with any known hypersensitivity to EC-MPS or everolimus or other components of the formulation (e.g., lactose)
* Patients with a history of severe rejection (according to BANFF criteria) within 3 months of enrollment in this trial.
* Changes to the immunosuppressive regimen during the last 3 months due to immunologic reasons.
* Patients with thrombocytopenia (platelets <100,000/mm3), with an absolute neutrophil count of <1,500/mm3 and/or leukocytopenia (leukocytes <4,500/mm3), and/or hemoglobin <9.0 g/dL at baseline.
* Patients with proteinuria at baseline (> 1g/d)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2004-01; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Kinetic Profiles (MPA, everolimus, and optional IMPDH) will be measured at day 0, 7 and 7 days after complete removal of CsA and last dose adjustment of everolimus due to trough level outside target range | 7 days
Everolimus trough level will be measured at day 7, 14, 21, 28 and month 2, 4, 6, 9, 12 | 1 year

SECONDARY OUTCOMES:
Safety and tolerability of the treatment regimen consisting over a one year period | 1 year
Renal function during the course of the trial, especially after CNI withdrawal. | 1 year
Routine laboratory parameters during the course of the trial. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Klemens Budde, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité-Universitätsmedizin, Berlin, Germany